CLINICAL TRIAL: NCT00097773
Title: Effectiveness and Safety of Intermittent Antimicrobial Therapy for the Treatment of New Onset Pseudomonas Aeruginosa Airway Infection in Young Patients With Cystic Fibrosis
Brief Title: Comparison of Two Treatment Regimens to Reduce PA Infection in Children With Cystic Fibrosis
Acronym: EPIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other); CF Therapeutics Development Network Coordinating Center (Network)
Responsible Party: Principal Investigator, Bonnie Ramsey, Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 169; U01HL080310 (NIH)
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive
Keywords: Lung Diseases; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Inhalation; Tobramycin; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cycled TOBI & placebo (Placebo Comparator): Tobramycin inhalation solution and oral placebo for six consecutive quarterly cycles
  Interventions: Drug: Tobramycin solution for inhalation (TOBI); Drug: Oral placebo
- Cycled TOBI & oral ciprofloxacin (Active Comparator): Tobramycin solution for inhalation and oral ciprofloxacin for six consecutive quarterly cycles.
  Interventions: Drug: Tobramycin solution for inhalation (TOBI); Drug: Oral ciprofloxacin
- Culture based TOBI & placebo (Placebo Comparator): Tobramycin solution for inhalation and oral placebo administered only when quarterly respiratory cultures are found positive for Pa.
  Interventions: Drug: Tobramycin solution for inhalation (TOBI); Drug: Oral placebo
- Culture based TOBI & oral cipro (Active Comparator): Tobramycin solution for inhalation and oral ciprofloxacin administered only when quarterly respiratory cultures are found positive for Pa.
  Interventions: Drug: Tobramycin solution for inhalation (TOBI); Drug: Oral ciprofloxacin

INTERVENTIONS:
Drug: Tobramycin solution for inhalation (TOBI) — Tobramycin solution for inhalation, 300 mg, administered twice daily for 28 days administered only when quarterly respiratory cultures are found positive for Pa.
  Other Names: TOBI, TIS
Drug: Oral placebo — Oral placebo for six consecutive quarterly cycles. For the initial 14 days of the 28-day treatment period, the participants will receive placebo, twice daily.
  Other Names: Placebo
  Arms: Culture based TOBI & placebo; Cycled TOBI & placebo
Drug: Oral ciprofloxacin — Oral ciprofloxacin for six consecutive quarterly cycles. For the initial 14 days of the 28-day treatment period, the participants will receive oral ciprofloxacin, 15-20 mg/kg/dose, twice daily.
  Other Names: Cipro; Ciprofloxacin
  Arms: Culture based TOBI & oral cipro; Cycled TOBI & oral ciprofloxacin

SUMMARY:
Cystic fibrosis (CF) is a chronic disease that significantly affects an individual's lung function. Antibiotic medications have been proven effective at reducing Pseudomonas aeruginosa (PA) infection, which is one of the main causes of death in individuals with CF. The purpose of this study is to compare the effectiveness of treatment based on quarterly culture results versus consistent quarterly antibiotic treatment at reducing PA infection in children with CF.

DETAILED DESCRIPTION:
CF is an inherited disease that causes mucus to build up in the lungs and digestive tract, which can cause lung infections and digestive problems. It is the most common type of chronic lung disease in children and young adults and may result in early death. There is no cure for this disease. The primary cause of death in individuals with CF is progressive obstructive pulmonary disease associated with chronic Pseudomonas aeruginosa (PA) infection. PA infection can occur early in life and can become highly resistant to antibiotics. Once an individual has been diagnosed with chronic PA infection, it is almost impossible to manage effectively. The need exists for an effective treatment to control and eliminate PA infection. Past research has shown that if PA infection is treated early, there is a greater likelihood that it may be eliminated completely. This study will examine two treatment regimens to compare which is more effective at eliminating PA infection. In the first regimen, participants will receive antibiotic treatment at various times throughout the study, based on findings of PA respiratory cultures obtained on a quarterly basis. In the second regimen, participants will receive antibiotic medications in consistent, quarterly cycles throughout the study. The antibiotic medications used in this study will be ciprofloxacin and inhaled tobramycin, which will be administered with a nebulizer. Both of these medications have been proven effective at treating bacterial lung infections. The overall purpose of this study is to compare the effectiveness of culture-based treatment versus consistent treatment at reducing PA infection in children with CF.

This 18-month study will enroll children with CF. For the first 28 days of the study, all participants will receive inhaled tobramycin. For the initial 14 days of this 28-day period, half of the participants will also receive either ciprofloxacin or placebo. If respiratory cultures after three weeks of treatment confirm the presence of PA, participants will receive tobramycin for an additional 28 days. Participants will then be randomly assigned to one of four treatment options: tobramycin and placebo for six consecutive quarterly cycles; tobramycin and ciprofloxacin for six consecutive quarterly cycles; tobramycin and placebo only when PA is found during quarterly respiratory cultures; or tobramycin and ciprofloxacin only when PA is found during quarterly respiratory cultures.

At the first study visit, participants will undergo a physical examination, a chest x-ray, and a review of their medical history. Lung function will be measured via spirometry (in children greater than four years of age who are able to perform spirometry), and hearing ability will be measured via audiometry (at selected sites). Blood will be drawn for laboratory tests, and a specimen will be obtained for a respiratory culture. Subsequent study visits will take place at Day 21, Weeks 10, 22, 34, 46, 58, and 70. At each visit, participants will undergo a physical examination and a spirometry test (as appropriate), and a respiratory specimen for PA culture and blood will again be collected. Participants will be required to maintain a medication diary throughout the study, and they will be contacted between visits to review medication adherence and test results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF, as determined by the 1997 CF Consensus Conference criteria: sweat chloride level greater than 60 milliequivalent/liter (mEq/L) by quantitative pilocarpine iontophoresis; or a genotype with two identifiable mutations consistent with CF; or an abnormal nasal transepithelial potential difference and one or more clinical features consistent with CF
* For participants greater than 15 months of age: documented new onset of positive oropharyngeal, sputum, or lower respiratory tract culture for PA within 6 months of study entry, defined as either: 1) first lifetime documented PA positive culture; or 2) PA recovered after at least a 2-year history of PA negative respiratory cultures (at least one culture per year)
* For participants 12-15 months of age: at least one documented positive oropharyngeal, sputum, or lower respiratory tract culture for PA since birth or CF diagnosis
* Clinically stable with no evidence of any significant respiratory symptoms or chest radiograph findings at screening that would require administration of intravenous anti-pseudomonal antibiotics, oxygen supplementation, or hospitalization

Exclusion Criteria:

* History of aminoglycoside hypersensitivity or adverse reaction to inhaled aminoglycoside
* History of hypersensitivity or adverse reaction to ciprofloxacin or other fluoroquinolone medications
* History of persistent, unresolved hearing loss documented by audiometric testing on at least two occasions and not associated with middle ear disease or an abnormal tympanogram
* Abnormal kidney function at study entry (defined as a serum creatinine level greater than 1.5 times the upper limit of normal for participant's age)
* Abnormal liver function test results at study entry (defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels greater than two times the upper limit of normal range)
* Use of any investigational drug within 30 days of study entry
* Use of loop diuretics, phenytoin, warfarin, theophylline, or other methylxanthines within 30 days of study entry
* Use of more than one course of intravenous anti-pseudomonal antibiotics (at least 10 continuous days of medication use) or more than one course of inhaled anti-pseudomonal antibiotics (at least 28 continuous days of medication use) within 2 years of study entry; intravenous or inhaled anti-pseudomonal antibiotics must be stopped at least 30 days prior to study entry
* Chronic macrolide use (more than 90 day duration) in the 3 months prior to study entry
* Presence of a condition or abnormality that would compromise the participant's safety or the quality of the study data, in the opinion of the investigator

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie W. Ramsey, Principal Investigator — University of Washington; George Retsch-Bogart, MD, Principal Investigator — University of North Carolina, Chapel Hill; Miriam Treggiari, MD, Principal Investigator — University of Washington
Locations (54):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Northern California Kaiser Cystic Fibrosis Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Denver, Aurora, Colorado
  - duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital Cystic Fibrosis Center, St. Petersburg, Florida
  - Emory University Cystic Fibrosis Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital/Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Spectrum Health Hospitals - DeVos Children's, Grand Rapids, Michigan
  - Children's Hospitals & Clinics, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Albany Medical College, Albany, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Children's Hospital, Columbus, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Children's Hospital at Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital & Regional Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Treggiari MM, Rosenfeld M, Mayer-Hamblett N, Retsch-Bogart G, Gibson RL, Williams J, Emerson J, Kronmal RA, Ramsey BW; EPIC Study Group. Early anti-pseudomonal acquisition in young patients with cystic fibrosis: rationale and design of the EPIC clinical trial and observational study'. Contemp Clin Trials. 2009 May;30(3):256-68. doi: 10.1016/j.cct.2009.01.003. Epub 2009 Jan 15. PMID 19470318
- [Result] Treggiari MM, Retsch-Bogart G, Mayer-Hamblett N, Khan U, Kulich M, Kronmal R, Williams J, Hiatt P, Gibson RL, Spencer T, Orenstein D, Chatfield BA, Froh DK, Burns JL, Rosenfeld M, Ramsey BW; Early Pseudomonas Infection Control (EPIC) Investigators. Comparative efficacy and safety of 4 randomized regimens to treat early Pseudomonas aeruginosa infection in children with cystic fibrosis. Arch Pediatr Adolesc Med. 2011 Sep;165(9):847-56. doi: 10.1001/archpediatrics.2011.136. PMID 21893650
- [Derived] Sanders DB, Emerson J, Ren CL, Schechter MS, Gibson RL, Morgan W, Rosenfeld M; EPIC Study Group. Early Childhood Risk Factors for Decreased FEV1 at Age Six to Seven Years in Young Children with Cystic Fibrosis. Ann Am Thorac Soc. 2015 Aug;12(8):1170-6. doi: 10.1513/AnnalsATS.201504-198OC. PMID 26288390
- [Derived] Mayer-Hamblett N, Kloster M, Rosenfeld M, Gibson RL, Retsch-Bogart GZ, Emerson J, Thompson V, Ramsey BW. Impact of Sustained Eradication of New Pseudomonas aeruginosa Infection on Long-term Outcomes in Cystic Fibrosis. Clin Infect Dis. 2015 Sep 1;61(5):707-15. doi: 10.1093/cid/civ377. Epub 2015 May 13. PMID 25972024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from December 2004 to June 2009 from 55 Cystic Fibrosis Foundation accredited clinical centers throughout the US
Groups:
- Cycled TOBI and Oral Placebo: Tobramycin solution for inhalation (TOBI) and oral placebo for six consecutive quarterly cycles
- Cycled TOBI and Oral Ciprofloxacin: Tobramycin solution for inhalation (TOBI) and oral ciprofloxacin for six consecutive quarterly cycles
- Culture-Based TOBI and Oral Ciprofloxacin: Tobramycin solution for inhalation (TOBI) and oral ciprofloxacin administered only when quarterly respiratory cultures are found positive for Pseudomonas aeruginosa (Pa)
- Culture-Based TOBI and Oral Placebo: Tobramycin solution for inhalation (TOBI) and oral placebo administered only when quarterly respiratory cultures are found positive for Pseudomonas aeruginosa (Pa)
Period: Overall Study
Arm/Group | Cycled TOBI and Oral Placebo | Cycled TOBI and Oral Ciprofloxacin | Culture-Based TOBI and Oral Ciprofloxacin | Culture-Based TOBI and Oral Placebo
Started | 76 | 76 | 76 | 76
Completed | 68 | 68 | 68 | 73
Not Completed | 8 | 8 | 8 | 3
Not completed — Lost to Follow-up | 2 | 2 | 0 | 1
Not completed — Physician Decision | 2 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Groups:
- Cycled TIS w/Placebo: TOBI and oral placebo for six consecutive quarterly cycles
- Cycled TIS w/Cipro: TOBI and oral ciprofloxacin for six consecutive quarterly cycles
- Culture-Based TIS w/Placebo: TOBI and oral placebo administered only when quarterly respiratory cultures are found positive for Pseudomonas aeruginosa (Pa)
- Culture-Based TIS w/Cipro: TOBI and oral ciprofloxacin administered only when quarterly respiratory cultures are found positive for Pseudomonas aeruginosa (Pa)
- Total: Total of all reporting groups
Arm/Group | Cycled TIS w/Placebo | Cycled TIS w/Cipro | Culture-Based TIS w/Placebo | Culture-Based TIS w/Cipro | Total
Number analyzed (Participants) | 76 | 76 | 76 | 76 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76 | 76 | 76 | 76 | 304
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (3.43) | 5.9 (3.28) | 6.0 (3.74) | 5.0 (3.58) | 5.7 (3.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 32 | 40 | 37 | 154
  Male | 31 | 44 | 36 | 39 | 150
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 76 | 76 | 304

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pulmonary Exacerbation Requiring IV Antibiotics or Hospitalization
Description: The primary comparison is between the pooled culture-based group and the pooled cycled group. A secondary comparison is between the pooled ciprofloxacin group vs the pooled placebo group. Descriptive results are provided for the pooled treatment groups.
  Participants are represented once in the cycled and culture-based therapy columns, and once in the cipro and placebo columns.
Time Frame: Measured over the 18 month study
Population: Intent to treat
Measure: Number; unit: number of participants
Groups:
- Cycled TIS: Pooled Cycled tobramycin solution for inhalation (TIS) therapy group
- Culture-Based TIS: Pooled Culture-Based TIS therapy group
- Oral Ciprofloxacin: Pooled oral cipro group
- Oral Placebo: Pooled oral placebo group
Arm/Group | Cycled TIS | Culture-Based TIS | Oral Ciprofloxacin | Oral Placebo
Number analyzed (Participants) | 152 | 152 | 152 | 152
number of participants | 24 | 26 | 29 | 21
Statistical Analysis 1: Comparison: Cycled TIS vs Culture-Based TIS; The primary analysis compared the pooled Cycled Therapy group (n=152) vs. the Pooled culture-based therapy group (n=152). The null hypothesis was no difference between groups in the risk of pulmonary exacerbation requiring IV antibiotics or hospitalization. Assuming a total sample size of 300 (150 per group), the study provided 80% power to detect at least a 40% reduction in the risk of exacerbation in the cycled group as compared to the culture-based group at the two-sided alpha level of 5%; Test type: Superiority or Other; p = 0.86, Regression, Cox — There was no significant interaction with ciprofloxacin in this analysis; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.54 to 1.66] — risk of exacerbation comparing cycled therapy to culture-based therapy
Statistical Analysis 2: Comparison: Oral Ciprofloxacin vs Oral Placebo; A secondary comparison was between the pooled oral cipro (n=152)and pooled placebo groups (n=152. Null hypothesis was no difference between groups; Test type: Superiority or Other; p = 0.20, Regression, Cox; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.82 to 2.54] — risk of exacerbation comparing oral cipro to oral placebo

2. Secondary Outcome: Proportion of Participants With a Pa Positive Culture
Description: Proportion of participants with a Pa positive culture compared between (1) the pooled cycled therapy group (n=152) and pooled culture-based therapy group (n=152), and (2) between the pooled oral placebo (n=152)and pooled cipro groups (n=152).
  Participants are included once in the cycled and culture-based columns, and once in the oral cipro and placebo columns
Time Frame: Week 10 (after initial treatment course for Pa) through Month 18
Population: Intent to treat
Measure: Number; unit: Participants
Groups:
- Cycled TIS: Pooled Cycled TIS group
- Culture-Based TIS: Pooled Culture-Based TIS group
- Oral Cipro: Pooled oral cipro group
Arm/Group | Cycled TIS | Culture-Based TIS | Oral Cipro | Oral Placebo
Number analyzed (Participants) | 152 | 152 | 152 | 152
Participants
  No Pa positive cultures | 109 | 85 | 97 | 97
  1 Pa positive culture | 17 | 38 | 22 | 33
  2 Pa positive cultures | 9 | 18 | 13 | 14
  3 or more Pa positive cultures | 13 | 9 | 14 | 8
  Missing | 4 | 2 | 6 | 0
Statistical Analysis 1: Comparison: Cycled TIS vs Culture-Based TIS; Null hypothesis is that there is no difference between pooled cycled and culture-based treatment groups in the odds of a Pa positive culture over the 18 month study; Test type: Superiority or Other; p = 0.28, Regression, Logistic; No interaction with ciprofloxacin usage was observed; Odds Ratio (OR) = 0.78, 95% CI [0.49 to 1.23] — odds of a positive culture comparing cycled therapy to culture-based therapy
Statistical Analysis 2: Comparison: Oral Cipro vs Oral Placebo; Null hypothesis is that there is no difference between pooled cipro and placebo treatment groups in the odds of a Pa positive culture over the 18 month study; Test type: Superiority or Other; p = 0.67, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.71 to 1.71] — odds of a positive culture comparing the cipro group to the placebo group

3. Secondary Outcome: Number of Participants With a Pulmonary Exacerbation Requiring Oral, Inhaled, or Oral Antibiotics
Description: The primary comparison is between the pooled culture-based group and the pooled cycled group. No interactions with ciprofloxacin were identified. A secondary comparison is between the pooled ciprofloxacin group vs the pooled placebo group. Descriptive results are provided for the pooled treatment groups.
  Participants are represented once in the cycled and culture-based therapy columns, and once in the cipro and placebo columns.
Time Frame: Measured over the 18 month time period
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- Cycled TIS: Pooled Cycled TIS therapy group
Arm/Group | Cycled TIS | Culture-Based TIS | Oral Ciprofloxacin | Oral Placebo
Number analyzed (Participants) | 152 | 152 | 152 | 152
participants | 70 | 81 | 83 | 68
Statistical Analysis 1: Comparison: Cycled TIS vs Culture-Based TIS; The analysis compared the pooled Cycled Therapy group (n=152) vs. the Pooled culture-based therapy group (n=152). The null hypothesis was no difference between groups in the risk of pulmonary exacerbation; Test type: Superiority or Other; p = 0.18, Regression, Cox; No interaction with ciprofloxacin usage was observed; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.11] — Hazard ratio comparing cycled to culture based therapy
Statistical Analysis 2: Comparison: Oral Ciprofloxacin vs Oral Placebo; This analysis was between the pooled oral cipro (n=152)and pooled placebo groups (n=152. Null hypothesis was no difference between groups; Test type: Superiority or Other; p = 0.12, Regression, Cox; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.94 to 1.78] — Hazard ratio comparing cipro to placebo

ADVERSE EVENTS:
Time Frame: Randomization through Month 18
Groups:
- Culture-Based TIS w/Cipro: TOBI and oral ciprofloxacin administered only when quarterly respiratory cultures are found positive for PA
Arm/Group | Cycled TIS w/Placebo | Cycled TIS w/Cipro | Culture-Based TIS w/Placebo | Culture-Based TIS w/Cipro
Serious Adverse Events (participants affected / at risk) | 18/76 | 21/76 | 17/76 | 27/76
Other Adverse Events (participants affected / at risk) | 65/76 | 67/76 | 65/76 | 73/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycled TIS w/Placebo (N=76) | Cycled TIS w/Cipro (N=76) | Culture-Based TIS w/Placebo (N=76) | Culture-Based TIS w/Cipro (N=76)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Distal Intestinal Obstruction Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pseudomonas Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forced Expiratory Volume Decreased (Investigations) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Pulmonary Function Test Decreased (Investigations) | 3 (3) | 2 (3) | 1 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (9) | 2 (2) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenotonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central Venous Catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Tube Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrostomy Tube Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vesicoureteral Reflux Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycled TIS w/Placebo (N=76) | Cycled TIS w/Cipro (N=76) | Culture-Based TIS w/Placebo (N=76) | Culture-Based TIS w/Cipro (N=76)
Lymphadenopathy (Blood and lymphatic system disorders) | 12 (13) | 8 (8) | 13 (14) | 11 (12)
Ear Pain (Ear and labyrinth disorders) | 8 (13) | 9 (11) | 11 (18) | 17 (19)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 6 (6) | 10 (10) | 4 (5)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 4 (5) | 4 (4) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 7 (8) | 5 (8) | 4 (4) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 4 (7)
Abdominal Pain (Gastrointestinal disorders) | 17 (20) | 12 (15) | 16 (21) | 12 (15)
Abdominal Pain Upper (Gastrointestinal disorders) | 14 (22) | 18 (34) | 15 (35) | 17 (30)
Constipation (Gastrointestinal disorders) | 6 (8) | 9 (15) | 13 (14) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 15 (24) | 22 (40) | 22 (24) | 26 (49)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 5 (6)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 12 (21) | 6 (7) | 7 (11)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Post-Tussive Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Teething (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (52) | 30 (52) | 35 (49) | 37 (70)
Asthenia (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Chest Pain (General disorders) | 6 (8) | 7 (8) | 6 (8) | 11 (15)
Chills (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Crepitations (General disorders) | 0 (0) | 5 (6) | 0 (0) | 4 (4)
Exercise Tolerance Decreased (General disorders) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (19) | 7 (9) | 13 (21) | 10 (14)
Irritability (General disorders) | 4 (4) | 4 (5) | 0 (0) | 8 (11)
Pain (General disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 46 (85) | 45 (107) | 57 (138) | 57 (129)
Seasonal Allergy (Immune system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Conjunctivitis Infective (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Ear Infection (Infections and infestations) | 5 (6) | 12 (17) | 8 (8) | 17 (25)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (6) | 0 (0) | 0 (0) | 4 (6)
Otitis Media (Infections and infestations) | 17 (24) | 7 (7) | 21 (33) | 15 (23)
Pharyngitis Streptococcal (Infections and infestations) | 7 (10) | 9 (11) | 6 (9) | 11 (16)
Rhinitis (Infections and infestations) | 7 (10) | 10 (12) | 10 (11) | 6 (11)
Sinusitis (Infections and infestations) | 13 (20) | 13 (15) | 11 (16) | 22 (25)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 4 (4)
Arthropod Bite (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 5 (8) | 4 (5) | 6 (8)
Excoriation (Injury, poisoning and procedural complications) | 4 (5) | 4 (4) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 9 (13) | 10 (15) | 10 (13) | 8 (8)
Chest X-Ray Abnormal (Investigations) | 8 (8) | 7 (9) | 9 (9) | 8 (9)
Forced Expiratory Volume Decreased (Investigations) | 11 (16) | 12 (15) | 9 (10) | 9 (11)
Increased Anteroposterior Chest Diameter (Investigations) | 4 (4) | 5 (5) | 4 (5) | 0 (0)
Methicillin-Resistant Staphylococcal Aureus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pulmonary Function Test Decreased (Investigations) | 4 (5) | 5 (6) | 5 (5) | 9 (14)
Respiratory Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sputum Abnormal (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Weight Decreased (Investigations) | 7 (9) | 10 (12) | 6 (6) | 14 (17)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 17 (27) | 9 (10) | 9 (9) | 20 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17) | 14 (25) | 14 (18) | 12 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8) | 0 (0) | 5 (7)
Clubbing (Musculoskeletal and connective tissue disorders) | 7 (7) | 15 (16) | 7 (8) | 8 (9)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 6 (6) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 15 (27) | 10 (16) | 12 (14)
Dizziness (Nervous system disorders) | 0 (0) | 5 (7) | 6 (6) | 4 (7)
Headache (Nervous system disorders) | 38 (72) | 28 (69) | 24 (47) | 31 (75)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Decreased Activity (Psychiatric disorders) | 10 (11) | 5 (5) | 5 (5) | 7 (7)
Dysuria (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Bronchial Wall Thickening (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 62 (202) | 63 (240) | 65 (224) | 71 (282)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 16 (28) | 12 (26) | 15 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (9) | 13 (19) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (8) | 12 (20) | 8 (11)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 44 (88) | 38 (68) | 40 (85) | 48 (98)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (9) | 10 (12) | 6 (6)
Nasal Oedema (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (9) | 9 (11) | 12 (13)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9) | 9 (10) | 7 (7)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 19 (31) | 26 (51) | 24 (36) | 28 (59)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 23 (40) | 22 (38) | 28 (48)
Rales (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (19) | 11 (16) | 12 (16)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 17 (32) | 13 (15) | 13 (18)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 41 (100) | 48 (123) | 47 (119) | 50 (139)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 4 (4)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (6) | 0 (0) | 5 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (6) | 0 (0) | 5 (6)
Sputum Discolored (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (8) | 4 (4) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4) | 7 (7) | 5 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 15 (24) | 12 (16) | 17 (22)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (18)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (15) | 13 (18) | 16 (21) | 16 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Sinus Operation (Surgical and medical procedures) | 0 (0) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No